CLINICAL TRIAL: NCT07284732
Title: Effects of Pairing Transcutaneous Auricular Vagus Nerve Stimulation on Patients With Disorders of Consciousness: An Exploratory Single-Center Randomized Controlled Trial
Brief Title: Effect of taVNS on Patients With Disorders of Consciousness
Acronym: taVNS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Qiuyou Xie, principal investigator, Zhujiang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L20251010
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Disorders of Consciousness
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Closed-Loop transcutaneous auricular vagus nerve stimulation (Experimental): Stimulation will be delivered on the left cymba conchae using a silicone electrode
  Interventions: Device: transcutaneous auricular vagus nerve stimulation

INTERVENTIONS:
Device: transcutaneous auricular vagus nerve stimulation — The stimulation protocol consisted of pulse trains at a frequency of 100 Hz. A total of 400 paired RAVANS pulses were delivered per session. The intervention was administered twice daily for 10 consecutive days, resulting in a total of 20 sessions.

SUMMARY:
Consciousness disorders following severe brain injury refer to a series of disturbances in arousal and cognition secondary to organic brain diseases, including Unresponsive Wakefulness Syndrome (UWS) (also termed Vegetative State, VS) and Minimally Conscious State (MCS). DoC is listed in the International Statistical Classification of Diseases and Related Health Problems, though it is not currently recognized as an independent and consistent diagnostic category. According to epidemiological surveys, conservative estimates suggest that 70,000 to 100,000 new cases of DoC are reported annually in China, posing significant challenges for clinical diagnosis and treatment. Accurately assessing DoC, understanding its neurobiological underpinnings, and developing effective rehabilitation strategies remain subjects requiring further investigation through both clinical and basic neuroscience research.

Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) is a non-invasive brain stimulation technique that delivers electrical impulses to the auricular branch of the vagus nerve. Substantial evidence indicates that taVNS serves as a therapeutic intervention for various neurological and psychiatric disorders, such as epilepsy, treatment-resistant depression, migraines, and cognitive impairments. As an emerging neurostimulation technique, taVNS has been investigated for its potential to promote the recovery of awareness in patients with DoC. However, clinical evidence remains limited, underscoring the need for further trials to substantiate its efficacy. Developed from traditional implanted VNS, taVNS offers high safety and minimal to negligible side effects, presenting a promising therapeutic avenue for patients with severe traumatic brain injury and disorders of consciousness.

Methods: This study is a single-arm trial. A total of 20 patients are planned to be enrolled. Each patient will receive transcutaneous auricular vagus nerve stimulation (taVNS) twice daily over a period of 10 consecutive days, totaling 20 sessions. Primary and secondary outcome measures will be assessed at baseline and after the completion of taVNS treatment. The primary efficacy endpoint will be the change in behavioral responses as evaluated by the Coma Recovery Scale-Revised (CRS-R). Additionally, resting-state high-density electroencephalography (EEG) and combined transcranial magnetic stimulation with EEG (TMS-EEG) recordings will be utilized to investigate the neurophysiological correlates of taVNS intervention.

Discussion: This study will provide valuable insights to inform the selection of treatment approaches for patients with disorders of consciousness. By employing a pre-post within-subject comparison design, it aims to validate the therapeutic role of Closed-Loop Transcutaneous Auricular Vagus Nerve Stimulation (CL-taVNS) in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years, with a disease duration exceeding 28 days but not longer than 1 year.
* Patients diagnosed with disorders of consciousness (DoC), specifically classified as either vegetative state (VS) or minimally conscious state (MCS) according to the Coma Recovery Scale-Revised (CRS-R) based on international guidelines.
* No prior history of neuropsychiatric disorders.
* Absence of contraindications to transcutaneous auricular vagus nerve stimulation (taVNS) or electroencephalography (EEG), and no concurrent use of sedatives or medications that may interfere with cerebral stimulation-including Na⁺ or Ca²⁺ channel blockers or NMDA receptor antagonists.
* Intact skin at the auricular site.

Exclusion Criteria:

* Participation in other trials involving non-invasive or invasive neuromodulation.
* Uncontrolled epilepsy, defined as seizures occurring within 4 weeks prior to enrollment.
* Presence of cranial metal implants, pacemakers, craniotomy at the stimulation site, implanted brain devices, or similar conditions.
* Cardiac arrhythmia or other significant cardiovascular abnormalities;
* History of respiratory disorders, including dyspnea, asthma, or hyperventilation.
* History of vasovagal syncope.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline JKF Coma Recovery Scale-Revised(CRS-R) | immediately after 10 days TaVNS session
  The CRS-R comprises six subscales designed to assess auditory, visual, oromotor, communication,and arousal processes. Each CRS-R subscale score is determined based on the presence or absence of specific behavioral responses to sensory stimuli. The total score ranges from 0 to 23, with higher scores indicating a higher level of consciousness in patients with DoC.

SECONDARY OUTCOMES:
Change from Baseline Resting-State EEG | immediately after 10 days TaVNS session
  EEG data will be recorded for 10 minutes using a 66-channel cap arranged according to the International 10-20 System. From artifact-free EEG epochs, relative spectral power (RSP) and functional connectivity (FC) will be derived across five frequency bands: δ (1-4 Hz), θ (4-8 Hz), α (8-13 Hz), β (13-30 Hz), and γ (30-45 Hz). All analyses of RSP and FC will be performed offline.
Change from Baseline TMS-EEG | immediately after 10 days TaVNS session
  Transcranial magnetic stimulation combined with electroencephalography (TMS-EEG) is an effective way to measure cortical activity.In this study, PCIst, a derivative version of PCI, PCIst was chosen as an alternative, which estimates the complexity of TMS perturbations by signal decomposition and recurrence quantification analysis (RQA).

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No